CLINICAL TRIAL: NCT00909753
Title: A Single-Dose, Comparative Bioavailability Study of Two Formulations of Ursodiol 500 mg Tablets Under Fed Conditions
Brief Title: Ursodiol 500 mg Tablets Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2006-1284
Record Dates: First submitted 2009-05-26; First posted 2009-05-28 (Estimated); Results first posted 2009-07-21 (Estimated); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ursodiol (test) First (Experimental): Ursodiol Tablets, 500 mg
  Interventions: Drug: Ursodiol
- Urso Forte™ (reference) First (Active Comparator): Urso Forte™ Tablets, 500 mg
  Interventions: Drug: Urso Forte™

INTERVENTIONS:
Drug: Ursodiol — Ursodiol Tablets, 500 mg
  Arms: Ursodiol (test) First
Drug: Urso Forte™ — Urso Forte™ Tablets, 500 mg
  Arms: Urso Forte™ (reference) First

SUMMARY:
The objective of this study was to evaluate the comparative bioavailability between Ursodiol 500 mg Tablets (test) and Urso Forte™ 500 mg Tablets (reference)after a single-dose in healthy subjects under fed conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smoking male and female subjects, 18 years of age or older.
* BMI ≥ 19 and ≤ 30.
* Negative for:

  1. HIV.
  2. Hepatitis B surface antigen and Hepatitis C antibody.
  3. Using drugs of abuse test (marijuana, amphetamines, barbiturates, cocaine, opiates, benzodiazepines and methadone).
  4. Urine cotinine test
  5. Serum HCG consistent with pregnancy (females only)
* No significant diseases or clinically significant findings in a physical examination.
* No clinically significant abnormal laboratory values.
* No clinically significant findings in vital signs measurements and a 12-lead electrocardiogram (ECG).
* Be informed of the nature of the study and given written consent prior to receiving any study procedure.
* Females who participate in this study are:

  1. unable to have children (e.g. post-menopausal, tubal ligation, hysterectomy) OR
  2. willing to remain abstinent [not engage in sexual intercourse] OR
  3. willing to use an effective method of double-barrier birth control (e.g. partner using condom and female using diaphragm, contraceptive sponge, spermicide or IUD)
* Females who participate in this study are not pregnant and/or non-lactating.

Exclusion Criteria:

* Known history or presence of any clinically significant medical condition.
* Known or suspected carcinoma.
* Known history or presence of:

  1. Hypersensitivity or idiosyncratic reaction to ursodiol and/or any other drug substances with similar activity.
  2. Alcoholism within the last 12 months.
  3. Drug dependence and/or substance abuse.
  4. Use of tobacco or nicotine-containing products within the last 6 months.
* On a special diet within 4 weeks prior to drug administration (e.g. liquid, protein, raw food diet).
* Participated in another clinical trial or received and investigational product within 30 days prior to drug administration.
* Donated up to 250 mL of blood within the previous 30 days OR Donated from 251 to 499 mL of blood in the previous 45 days OR Donated more than 499 mL of blood in the previous 56 days (based on the Canadian Blood Services guideline for blood donation.
* Females taking oral or transdermal hormonal contraceptives within 14 days preceding period 1 dosing.
* Females having taken implanted or injected hormonal contraceptives within 6 months prior to period 1 dosing.
* Requirement of any non-topical medication (prescription and/or over-the-counter, with systemic absorption) on a routine basis.
* Difficulty fasting or consuming the standard meals.
* Do not tolerate venipuncture.
* Unable to read or sign the ICF.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2006-09; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xueyu (Eric) Chen, MD, PhD, FRCP(C), Principal Investigator — Pharma Medica Research, Inc.
Locations (1):
- Pharma Medica Research Inc., Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Ursodiol (Test) First: Ursodiol Tablets, 500 mg (test) dosed in first period followed by UrsoForte™ Tablets, 500 mg (reference) dosed in second period.
- Urso Forte™ (Reference) First: Urso Forte™ Tablets, 500 mg (reference) dosed in first period followed by Ursodiol Tablets, 500 mg (test) dosed in second period.
Period: Period: First Intervention
Arm/Group | Ursodiol (Test) First | Urso Forte™ (Reference) First
Started | 46 | 46
Completed | 46 | 46
Not Completed | 0 | 0
Period: Period: Washout of 28 Days
Arm/Group | Ursodiol (Test) First | Urso Forte™ (Reference) First
Started | 46 | 46
Completed | 44 | 43
Not Completed | 2 | 3
Not completed — Protocol Violation | 2 | 3
Period: Period: Second Intervention
Arm/Group | Ursodiol (Test) First | Urso Forte™ (Reference) First
Started | 44 | 43
Completed | 43 | 43
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ursodiol (Test) First | Urso Forte™ (Reference) First | Total
Number analyzed (Participants) | 46 | 46 | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 46 | 92
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 17 | 30
  Male | 33 | 29 | 62
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 31 | 33 | 64
  Black | 13 | 11 | 24
  Asian | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  Canada | 46 | 46 | 92

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Concentration - for Total Ursodiol
Description: Bioequivalence based on Cmax
Time Frame: Blood samples collected over 72 hour period
Population: Data from all subjects who completed the study was included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Ursodiol: Ursodiol Tablets, 500 mg dosed in either period
- Urso Forte™: Urso Forte™ Tablets, 500 mg dosed in either period
Arm/Group | Ursodiol | Urso Forte™
Number analyzed (Participants) | 86 | 86
ng/mL | 6763.805 (2305.341) | 7461.161 (2922.024)
Statistical Analysis 1: Comparison: Ursodiol vs Urso Forte™; Test type: Non-Inferiority or Equivalence — Analysis of Variance (ANOVA) will be applied to log-transformed AUC and Cmax parameters; Geometric Test/Ref Ratio x 100 = 92.5, 90% CI [85.8 to 99.7] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

2. Primary Outcome: AUC0-72 - Area Under the Concentration-time Curve From Time Zero to 72 Hours Post Dose - for Total Ursodiol
Description: Bioequivalence based on AUC0-72
Time Frame: Blood samples collected over 72 hour period
Population: Data from all subjects who completed the study was included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Ursodiol | Urso Forte™
Number analyzed (Participants) | 86 | 86
ng*h/mL | 84789.776 (33376.080) | 87925.305 (30085.315)
Statistical Analysis 1: Comparison: Ursodiol vs Urso Forte™; Test type: Non-Inferiority or Equivalence — Analysis of Variance (ANOVA) will be applied to log-transformed AUC and Cmax parameters; Geometric Test/Ref Ratio x 100 = 95.5, 90% CI [92.2 to 98.9] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

3. Primary Outcome: Cmax for Unconjugated Ursodiol
Description: Bioequivalence based on Cmax
Time Frame: Blood samples collected over 72 hour period
Population: Data from all subjects who completed the study was included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ursodiol | Urso Forte™
Number analyzed (Participants) | 86 | 86
ng/mL | 5818.644 (2145.519) | 6549.897 (2681.097)
Statistical Analysis 1: Comparison: Ursodiol vs Urso Forte™; Test type: Non-Inferiority or Equivalence — Analysis of Variance (ANOVA) will be applied to log-transformed AUC and Cmax parameters; Geometric Test/Ref Ratio x 100 = 90.4, 90% CI [83.1 to 98.3] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

4. Primary Outcome: AUC0-72 for Unconjugated Ursodiol
Description: Bioequivalence based on AUC0-72
Time Frame: Blood samples collected over 72 hour period
Population: Data from all subjects who completed the study was included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Ursodiol | Urso Forte™
Number analyzed (Participants) | 86 | 86
ng*h/mL | 28543.339 (21022.046) | 30951.831 (16492.541)
Statistical Analysis 1: Comparison: Ursodiol vs Urso Forte™; Test type: Non-Inferiority or Equivalence — Analysis of Variance (ANOVA) will be applied to log-transformed AUC and Cmax parameters; Geometric Test/Ref Ratio x 100 = 90.5, 90% CI [85.5 to 95.9] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

5. Primary Outcome: Cmax for Total Ursodiol - Baseline Corrected
Description: Bioequivalence based on Cmax
Time Frame: Blood samples collected over 72 hour period
Population: Data from all subjects who completed the study was included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ursodiol | Urso Forte™
Number analyzed (Participants) | 86 | 86
ng/mL | 6659.969 (2304.322) | 7363.215 (2899.526)
Statistical Analysis 1: Comparison: Ursodiol vs Urso Forte™; Test type: Non-Inferiority or Equivalence — Analysis of Variance (ANOVA) will be applied to log-transformed AUC and Cmax parameters; Geometric Test/Ref Ratio x 100 = 92.2, 90% CI [85.5 to 99.5] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

6. Primary Outcome: AUC0-72 for Total Ursodiol - Baseline Corrected
Description: Bioequivalence based on AUC0-72
Time Frame: Blood samples collected over 72 hour period
Population: Data from all subjects who completed the study was included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Ursodiol | Urso Forte™
Number analyzed (Participants) | 86 | 86
ng*h/mL | 77392.805 (25146.096) | 80992.000 (22688.058)
Statistical Analysis 1: Comparison: Ursodiol vs Urso Forte™; Test type: Non-Inferiority or Equivalence — Analysis of Variance (ANOVA) will be applied to log-transformed AUC and Cmax parameters; Geometric Test/Ref Ratio x 100 = 95.0, 90% CI [91.3 to 98.7] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

7. Primary Outcome: Cmax for Unconjugated Ursodiol - Baseline Corrected
Description: Bioequivalence based on Cmax
Time Frame: Blood samples collected over 72 hour period
Population: Data from all subjects who completed the study was included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ursodiol | Urso Forte™
Number analyzed (Participants) | 86 | 86
ng/mL | 5794.876 (2147.270) | 6522.456 (2679.132)
Statistical Analysis 1: Comparison: Ursodiol vs Urso Forte™; Test type: Non-Inferiority or Equivalence — Analysis of Variance (ANOVA) will be applied to log-transformed AUC and Cmax parameters; Geometric Test/Ref Ratio x 100 = 90.4, 90% CI [83.1 to 98.3] — Bioequivalence is established when 90% COnfidence Interval falls within 80-125

8. Primary Outcome: AUC0-72 for Unconjugated Ursodiol - Baseline Corrected
Description: Bioequivalence based on AUC0-72
Time Frame: Blood samples collected over 72 hour period
Population: Data from all subjects who completed the study was included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Ursodiol | Urso Forte™
Number analyzed (Participants) | 86 | 86
ng*h/mL | 26921.471 (17284.940) | 29177.523 (12620.441)
Statistical Analysis 1: Comparison: Ursodiol vs Urso Forte™; Test type: Non-Inferiority or Equivalence — Analysis of Variance (ANOVA) will be applied to log-transformed AUC and Cmax parameters; Geometric Test/Ref Ratio x 100 = 90.5, 90% CI [85.0 to 96.3] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator is not allowed to discuss or publish trial results.